CLINICAL TRIAL: NCT00111995
Title: A Randomized, Double-Blind Study Comparing Aranesp® (Darbepoetin Alfa) and Recombinant Human Erythropoietin (rHuEPO) in the Treatment of Anemia in African-American Subjects With Chronic Renal Failure (CRF) Receiving Hemodialysis
Brief Title: Evaluating Aranesp® for the Treatment of Anemia in African-American Subjects With Chronic Renal Failure (CRF) Receiving Hemodialysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 20010125
Record Dates: First submitted 2005-05-27; First posted 2005-05-30 (Estimated); Last update posted 2008-08-08 (Estimated); Status verified 2008-08

CONDITIONS: Chronic Renal Failure; Anemia
Keywords: Chronic Renal Failure (CRF); Anemia
MeSH Terms: conditions — Kidney Failure, Chronic; Anemia | interventions — Darbepoetin alfa

INTERVENTIONS:
Drug: Aranesp®

SUMMARY:
This study is designed to evaluate the hemoglobin response to Aranesp® (darbepoetin alfa) in black subjects (African-Americans) with chronic renal failure (CRF) receiving hemodialysis and to examine the safety profile.

ELIGIBILITY:
Inclusion Criteria: - Diagnosis of CRF and 3 times weekly prescribed hemodialysis treatments for at least 8 weeks before signing informed consent - No planned change in dialysis modality or schedule - Black (as indicated on the Chronic Medical Evidence Disease Report, CMMS Form 2728) - Hemoglobin 9.5 to 12.5 g/dL on 2 consecutive occasions during the screening period (1 week + 2 days apart) and baseline hemoglobin level of 9.5 - 12.5 g/dL (defined as the mean of all measurements taken during the screening and baseline periods) - Transferrin saturation greater than or equal to 20% but less than or equal to 50% - Stable rHuEPO therapy given 3 times per week by intravenous (IV) route of administration for 6 weeks before randomization (stable is defined as less than or equal to 25% change in prescribed dose over 6 weeks, same route of administration, and no more than 1 missed or withheld dose during each of the two 3-week periods before randomization) Exclusion Criteria: - Scheduled for a living-related or living non-related donor transplant - rHuEPO dose greater than 40,000 units weekly - Uncontrolled hypertension (postdialysis diastolic blood pressure greater than 105 mmHg and/or systolic blood pressure greater than 180 mmHg on more than 1 occasion as noted in the collected blood pressure measurements during the screening/baseline period) - Congestive heart failure (New York Heart Association [NYHA] Class III or IV) - Major surgery (excluding vascular access surgery) within 8 weeks before signing informed consent and during screening/baseline - Clinical evidence of active inflammatory disease requiring cyclophosphamide, azathioprine, prednisone or other immunosuppressive therapy within 8 weeks before signing the informed consent and during screening/baseline - Currently (at the signing of the informed consent) receiving antibiotics for a systemic infection and during screening/baseline - Known positivity for HIV antibody or hepatitis B surface antigen - Grand mal seizures within the last year - Clinical evidence of current malignancy (other than non-melanomatous skin malignancy), and/or receiving chemotherapy, and/or radiation therapy for malignancies within 8 weeks of signing the informed consent and during screening/baseline - Active systemic hematologic disease (e.g., sickle cell anemia, myelodysplastic syndromes, hematological malignancy, myeloma, hemolytic anemia) within 8 weeks of signing the informed consent and during screening/baseline - Clinical evidence of severe hyperparathyroidism (parathyroid hormone [PTH] level greater than 1500 pg/mL or biopsy-proven bone marrow fibrosis) at last measurement - ALT or AST greater than 2x the upper limit of the normal range - Red blood cell transfusions within 8 weeks before signing the informed consent and during screening/baseline - Known hypersensitivity to human serum albumin (HSA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2002-05

PRIMARY OUTCOMES:
Mean hemoglobin level during the evaluation period

SECONDARY OUTCOMES:
The nature, frequency, severity, relationship to treatment, and outcome of adverse events with specific attention to hypertensive events

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_33_NESP_20010125.pdf
- See also: FDA-approved Drug Labeling — http://www.aranesp.com/